CLINICAL TRIAL: NCT02036606
Title: Psychopathological and Cognitive Mechanisms of Racing and Crowded Thoughts in Mood Disorders
Brief Title: Racing and Crowded Thoughts in Mood Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 5582
Record Dates: First submitted 2014-01-06; First posted 2014-01-15 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- mood disorders: Questionary and neuropsychological tasks will be administered
  Interventions: Behavioral: questionary
- control: Questionary and neuropsychological tasks will be administered
  Interventions: Behavioral: questionary

INTERVENTIONS:
Behavioral: questionary

SUMMARY:
Racing thoughts relate to subjective acceleration of thinking which has been essentially associated with manic episodes in bipolar disorder. Qualitatively, the phenomenology of racing thoughts in major depression seems to differ from rumination and pure manic racing thoughts: thoughts of all kinds accumulate in the patient's head. Recent qualitative evidence is consistent with the existence of these two kinds of "thought overactivity" related to mood disorders. In order to evaluate this and better understand the psychopathological and cognitive mechanisms that underlie thought overactivity in mood disorders, we have created a 34-item self-questionnaire - the Racing and Crowded Thoughts Questionnaire (RCTQ) and a number of neuropsychological tasks (time perception, cognitive flexibility). Also, given the relationship between mood disorders and creativity, it is likely that thought overactivity is related to increased creativity. We aim at evaluating this relationship through the French version of the Cognitive Processes Associated with Creativity scale (CPAC).

ELIGIBILITY:
Inclusion Criteria:

* Bipolar disorder or depressive disorder
* 18 -65 years old

Exclusion Criteria:

* neurological conditions or sequelae
* substance abuse in the last 10 months
* schizophrenia
* ADHD
* Borderline personality disorder
* Pregnant women- Subjects under legal supervision

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2014-04 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Validation of the scale of Crowded Racing Thoughts Questionary = (RCTQ scale that assesses the two forms of racing thoughts) | one week
  Demonstrated a two-factor structure (crowded and racing) assessment concurrent and discriminant validity.

SECONDARY OUTCOMES:
Evaluation of executive and temporal mechanisms involved in racing thoughts | one week

OTHER OUTCOMES:
Validation of the French version of the scale Cognitive Processes Associated with Creativity or CPAC scale (scale that assesses creativity) | one week

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Bertschy, PHDMD, Principal Investigator — Les Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de psychiatrie 2 , Les Hôpitaux Universitaires de Strasbourg, Strasbourg, Alsace, France